CLINICAL TRIAL: NCT05981859
Title: Safety and Efficacy of PCI Cardiac Mapping System Workstation 'AVIAR (MX-02)' in Patients Undergoing Percutaneous Coronary Intervention (PCI): Prospective, Multi-center, Single-arm, Open, Post-approval Clinical Trial
Brief Title: AVIAR(MX-02) Robotic-assisted Percutaneous Coronary Intervention
Acronym: RoboticPCI
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: LN Robotics (Unknown)
Responsible Party: Principal Investigator, Seung-Whan Lee, M.D., Ph.D., Principle Investigator, Asan Medical Center
Other Study IDs: 2023-0838
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Percutaneous Coronary Intervention
Keywords: Robotic PCI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of the steerable catheter control system 'AVIAR(MX-02)', which remotely controls the guidewire and stent/balloon during the percutaneous coronary intervention (PCI) for those who have suspected coronary artery disease (CAD) and need PCI (for product approval from the MFDS).

DETAILED DESCRIPTION:
The potential subjects who meet the "Coronary Angiography Selection/Exclusion Criteria" are eligible to be enrolled in the clinical trial. These individuals will undergo the standard pre-procedural preparations and receive local anesthesia on the day of the procedure. The angiography will be performed using the investigational medical device "AVIAR (MX-02)" via a percutaneous coronary intervention procedure. After the procedure, the subjects will remain in a supine position for approximately 4 hours in the recovery room or hospital room to ensure absolute stability. During this time, the investigator will observe the puncture site for hemostasis and monitor for any adverse events.

Within 2 days after the procedure or prior to discharge, the subjects will undergo safety assessments and evaluations for the occurrence of any adverse events or serious adverse events. Additionally, at the 1-month follow-up, all required follow-up tests will be completed, and if no adverse events have occurred or if any previously occurring adverse events have been resolved, the clinical trial for that particular subject will be concluded. However, if any adverse events remain unresolved and are deemed unrelated to the clinical trial by the investigator, the trial may be terminated for that subject.

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria:

  1. Adult women and men who are aged ≥19 and <75 years 2. Those who are suspected of stable angina and need percutaneous coronary intervention 3. Those who voluntarily decided to participate in this clinical trial and agreed in writing to the informed consent form 4. Those who are willing to comply with the protocol
* Angiographic Inclusion Criteria:

  1. If the lesion to be treated by coronary angiography (target lesion) is a native coronary artery lesion that has not been previously treated
  2. If the diameter of the lesioned vessel to be treated by coronary angiography (target vessel) is between 2.5 mm and 4.5 mm (by visual estimate).
  3. If diameter stenosis of the target vessel ≥50% (by visual estimate)

Exclusion Criteria:

* General Exclusion Criteria:

  1. Those with a left ventricular ejection fraction (LVEF) ≤ 30%
  2. Those who have a history of hypersensitivity to contrast agents such as stainless steel, cobalt-chromium, etc.
  3. Those who cannot stop taking antithrombotic drugs (anticoagulants, antiplatelet drugs)
  4. Those diagnosed with thrombocytopenia, thrombocytosis, neutropenia, or leukopenia
  5. Those who have a history of bleeding diathesis or coagulopathy or who refuse transfusion
  6. Those with a history of stroke (CVA) or transient ischemic attack (TIA) within 4 weeks from the screening date
  7. .Those with a history of active peptic ulcer or upper gastrointestinal bleeding within 24 weeks from the screening date
  8. Those with ST-elevation myocardial infarction (STEMI) (for example, those who started myocardial infarction symptoms within 72 hours from the screening date)
  9. Those with a history of cardiogenic shock or cardiac arrest
  10. Those who underwent coronary artery bypass grafting (CABG)
  11. Those who underwent percutaneous coronary intervention (PCI) within 72 hours from the screening date
  12. Those who had a major adverse coronary event (MACE) or a serious adverse event (SAE) after receiving the percutaneous coronary intervention (PCI) within 4 weeks from the screening date
  13. Those who are scheduled to undergo percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) within 4 weeks from the end of this clinical trial
  14. Those diagnosed with renal failure or those who are not suitable for angiography due to severe renal dysfunction (creatine > 2.0 mg/dL or eGFR (estimated glomerular filtration rate) < 30 ml/min) within one week prior to the date of coronary angiography
  15. Pregnant and breastfeeding women
  16. Women of childbearing potential who plan to become pregnant during this clinical trial
  17. A woman* or spouse who is likely to be pregnant does not agree to use contraception in a medically acceptable method of contraception** during the clinical trial

      * Pregnant women who have experienced first trimester (who have undergone surgical infertility (either uterine extraction or bilateral ovarian resection) or who have been defined as menopause for more than 12 months without any other reason are not women of childbearing age)
      * Hormonal contraception, vasectomy, intrauterine device (IUD) or IUS [intrauterine system], tubular ligation, double blocking (complex use of blocking methods such as condoms for men, condoms for women, cervical caps, contraceptive diaphragm, contraceptive sponge), and sanitizers a one-off method
  18. Those who are currently participating in other clinical trials or have experience participating in other clinical trials within 12 weeks from the screening date
  19. Other cases where the investigator determines that participation in a clinical trial is inappropriate ethically or because it may affect the study outcome.

      ☞The specific reason is recorded in the CRF
* Angiographic Exclusion Criteria:

  1. Those who require manual or mechanical thrombectomy, rotational atherectomy, directional coronary atherectomy (DCA), etc. in addition to stent placement and balloon dilatation
  2. If there are two or more target vessels
  3. If there are two or more target lesions in one blood vessel
  4. Any previous stent placement within 5 mm (proximal or distal) of the target lesion
  5. When the investigator determines that PCI is not suitable because the target lesion hasany of the following characteristics:

     * Is severely tortuous ≥45°

       * An ostial lesion in location ③The target vessel has evidence of intraluminal thrombus or severe tortuosity (> 90°) proximal to the target lesion ④Moderate or severe calcification at the target lesion or near the target lesion ⑤Target lesion that is located in a native vessel distal to an anastomosis with a saphenous vein graft or a left/right internal mammary artery (LIMA/RIMA) bypass and is approached through the by-pass graft ⑥If PCI cannot be performed for other reasons☞The specific reason is recorded in the CRF
  6. Unprotected left main coronary artery disease (an obstruction greater than 50% diameter stenosis in the left main coronary artery)
  7. If the investigator determines that the subject is not suitable for robotic-assisted PCI due to clinical and anatomical reasons.☞The specific reason is recorded in the CRF.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target number of participants for this clinical trial is a total of 20 patients during study duration . If subjects who meet the "Coronary Angiography Selection/Exclusion Criteria" are eligible to be enrolled in the clinical trial. These subjects will undergo the standard pre-procedural preparations and receive local anesthesia on the day of the procedure. The angiography will be performed using the investigational medical device "AVIAR (MX-02)" via a percutaneous coronary intervention procedure.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Clinical Success Criteria | 48hours
  If the residual stenosis rate of the lesion is less than 30% after completion of percutaneous coronary intervention using an investigational device If major adverse cardiovascular events (MACE)† have not occurred within 48 hours after the procedure or the time of discharge, whichever comes first
Technical Success Criteria | 48hours
  The stent (or balloon catheter) has successfully reached the target lesion without switching to manual manipulation
Effective dose(mSv) | 48hours
  The effective dose (mSv) is calculated as follows by multiplying the dose-length product (Dose-length product, DLP, mGy.cm) measured by the dosimeter on the chest of the subject and the operator and the weighting factor for each tissue
Procedure time (min) | 48hours
  - It is defined as the time from the manipulation of the guidewire using the investigational device to the removal of the guidewire.
  Total procedure time(min)
  - It is defined as the time from insertion of the arterial sheath to the point of removal of the sheath.

SECONDARY OUTCOMES:
TEAE | 1month
  treatment emergent adverse event, TEAE
MACE | 1month
  Major Adverse Cardiovascular Events) occurring in the study subjects during the clinical trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Whan Lee, MD, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - The Catholic University of Korea Eunpyeong St. Mary's Hospital, Seoul

REFERENCES:
- [Derived] Lee J, Kim TO, Lee PH, Kim YH, Kwon O, Lee SW. Safety and Feasibility of Robot-Assisted Percutaneous Coronary Intervention Using the AVIAR 2.0 System: A Prospective, Multi-Center, Single-Arm, Open, Investigator-Initiated, Post-Approval Clinical Trial. Korean Circ J. 2025 Apr;55(4):325-335. doi: 10.4070/kcj.2024.0226. Epub 2024 Nov 5. PMID 39733457